CLINICAL TRIAL: NCT06721364
Title: Validation and Testing of a Suicide Prevention Program in Improving the Mental Well-being of School-going Adolescents in Gilgit Baltistan, Pakistan: A Pre/Post-intervention Study Protocol
Brief Title: Validation and Testing of a Suicide Prevention Program to Improve Mental Well-Being Among Adolescents in Gilgit Baltistan, Pakistan: A Pre/Post-Intervention Protocol
Acronym: Protocol
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Yasmin Parpio, Principal, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ERC-2023-8509-24844; D43TW007292 (NIH)
Record Dates: First submitted 2024-10-20; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Suicide Prevention
Keywords: suicide prevention program; Strategies; intervention; measure; mental Wellbeing; Psychological health; Adolescent Health
MeSH Terms: conditions — Suicide Prevention; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention I:"RAAHI" RAAHI is a suicide literacy module that is specially designed to provide individuals with essential knowledge and skills by equipping them with tools to navigate the complexities of mental health and suicide prevention. This module aims to empower people to recognize signs of suicidal ideation, engage in empathetic communication through open discussion, combat stigma, and connect individuals in crisis with appropriate support and resources.
  Intervention II: "safeTALK" The &#34;safeTalk&#34; program is a psychoeducational initiative designed for suicide prevention among adolescents, consisting of a 4-hour workshop that incorporates presentations, videos, discussions, and questions.
Masking Description: Not any
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This is single arm pretest post-test, behavioural Suicide prevention intervention, so all the participants will be given the intervention
  Interventions: Behavioral: Suicide prevention treatment

INTERVENTIONS:
Behavioral: Suicide prevention treatment — Intervention I:"RAAHI" RAAHI is a suicide literacy module that is specially designed to provide individuals with essential knowledge and skills by equipping them with tools to navigate the complexities of mental health and suicide prevention. This module aims to empower people to recognize signs of suicidal ideation, engage in empathetic communication through open discussion, combat stigma, and connect individuals in crisis with appropriate support and resources. The duration of the module will be of three hours.
  Intervention II: "safeTALK" The "safeTalk" program is a psychoeducational initiative designed for suicide prevention among adolescents, consisting of a 4-hour workshop that incorporates presentations, videos, discussions, and questions.The workshop is designed according to the standard practices of safeTALK, to assist participants in (a) identifying warning signs of suicide; (b) Avoiding frequent impulses to overlook, dismiss, or avoid discussions about suicide.

SUMMARY:
Background Globally, around 800,000 people die annually by committing suicide with a disproportionate burden of 77% of these deaths occurring in low- and middle income countries. Suicidal ideation is frequently observed among adolescents and is directly associated with suicidal attempts. Pakistan has witnessed a marked escalation in suicide rates in recent years, with Gilgit-Baltistan reporting the highest incidence. Extensive scholarly inquiry suggests the potential role of suicide prevention strategies in mitigating suicidal ideation, attempts, and related fatalities. This study aims to validate and evaluate the efficacy of a locally contextualized suicide prevention programs called RAAHI (the Guide) and safeTALK in improving the mental wellbeing of school-going adolescents in the Gilgit Baltistan, Pakistan.

Method and Analysis The investigation will evaluate the effectiveness of a locally contextualized suicide prevention intervention program called RAAHI based on internationally tested out program named safeTALK among 267 adolescents attending 4 private schools in Gilgit Baltistan, Pakistan, followed by its contextual validation. 'RAAHI', a suicide literacy module is designed to equip individuals with the knowledge and skills to recognize signs of suicidal ideation, engage them empathetically, and connect those in crisis with support. It promotes open discussions, combats stigma, and encourages preventive measures for widespread suicide literacy. The, safeTalk a 4-hour psychoeducational workshop, aimed to prevent adolescent suicide through presentations, videos, discussions, and interactive sessions. Participants learned to identify warning signs, engage in TALK steps (Tell, Ask, Listen, KeepSafe), and connect individuals with crisis support.

Employing an & interrupted time-series design through a pre-post-test framework, the study will assess the impact of the intervention at various time points, post intervention (T2) and follow up after 8 weeks (T3). Descriptive and inferential analyses (paired t test, ANOVA) will be carried out to gauge alterations in each measured outcome (including knowledge, confidence, willingness, and help-seeking behaviors) during the course of the study.

Ethics and Dissemination The study protocol has been approved by the Ethical Review Committee of the Aga Khan University (registration number 2023-8509-24844). The study finding will be shared with the parents and school authorities through workshops conducted in Urdu. The study will be published in an open-access, peer-reviewed journal and presented at relevant conferences.

Strengths and Limitations

-Since there is no standard intervention available for suicide prevention for adolescents in Pakistani context, the current research will assist in up scaling contextualized suicide prevention intervention among school-going adolescents in Pakistan. However, due to time, budget and logistical constraints, this feasibility study will only be conducted In private schools of Gilgit Baltistan, Pakistan, limiting potentially diverse implementation experiences and outcomes in rural or public school settings. This may restrict the generalizability of the study findings. Moreover, employing a quasi-experimental design without an appropriate control group can potentially undermine the internal validity of the study.

DETAILED DESCRIPTION:
Introduction Suicide is a notable worldwide public health issue, resulting in a staggering number of fatalities annually (Milbourn et al., 2022). It ranks among the five leading causes of death, representing over one-third of all fatalities (Kinchin et al., 2020). The rising global suicide rate, surpassing 800,000 deaths annually, underscores the urgency of addressing this critical public health concern (WHO, 2024). In Australia, suicide is the leading cause of death among individuals aged 15-24 years, with an annual rate of 11.6 deaths per 100,000 population (Kinchin & Doran, 2018). Moreover, each suicide case potentially corresponds with over 20 attempted suicides, emphasizing the urgent need for suicide prevention interventions. WHO (2024) suggests an alarmingly high prevalence of suicidal ideation, encompassing non-fatal suicide attempts and self-harm. This tragic occurrence is widespread across the globe, with 77% of suicides taking place in low and middle-income countries (Kinchin et al., 2020).

Additionally, on a global scale, suicide is the fourth most common cause of mortality, for individuals between the ages of 15 and 29 (Organization, 2021). Over the past five years, the United Arab Emirates has recorded the highest rate of suicides globally, (11.4%), followed by the United Kingdom (10.80%), Nepal (10.33%), the United States of America (8.9%), and Pakistan (7%) (CDC, 2020). Within the spectrum of mental health disorders, suicide emerges as the foremost cause of violent death, even among the economically active age group of 15-44 years, (CDC, 2020). According to a meta-analysis, 22.3% of college students at some point in their lives had had suicidal thoughts, plans, or made attempt(Mortier et al., 2018). In addition, a survey of 8,113 high school students in Hawaii found that 16.4% of the adolescents reported having suicidal thoughts, and nearly 10% acknowledged having attempted suicide at least once in their lives (Ivey-Stephenson, 2020).

Adolescents are highly vulnerable to mental health problems due to academic stress, interpersonal issues, and the transition to adulthood; all these factors exert substantial influence on their physical, emotional, social, and mental well-being (Broad, Sandhu, Sunderji, & Charach, 2017). In Pakistan, these challenges are exacerbated by social and cultural pressures, mental health being considered as a stigma, and limited access to treatment, which impacts social functioning and academic success, with long-term consequences (Bibi, Blackwell, & Margraf, 2021).

Increasing evidence suggests that school-based suicide prevention interventions are effective in their approach (Kinchin et al., 2017). Such interventions span various levels of prevention, encompassing primary efforts, like public awareness campaigns; secondary approaches, such as gatekeeper training programs; tertiary interventions, like psychotherapy and postvention strategies, including survivor support groups.

Similarly, expanding the conventional classification of mental health interventions, suicide prevention strategies can be categorized into universal (targeting the general public) or selective (aimed at specific high-risk groups with elevated lifetime risk, such as adolescent and psychiatric inpatients) (Zalsman et al., 2016).

A meta-analysis of 13 RCTs found that the incidence of suicide-related behaviors among adolescents who participated in an educational program was significantly lower (31% reduction) than those in the control group (E. Bailey, Robinson, & Witt, 2023). Likewise, a review of 14 studies evaluating the effectiveness of school-based gatekeeper training programs found significant improvements in gatekeepers' understanding, perceptions, confidence, and willingness to take action. (Mo, Ko, & Xin, 2018).

A randomized controlled trial (RCT) of the Signs of Suicide (SOS) program found a significant reduction in suicide attempts among participants over a 3-month follow-up period (Schilling, Aseltine, & James, 2016). Moreover, a large-scale RCT of a Youth Aware of Mental Health (YAM) program, involving over 11,110 students from 10 European countries, showed a significant 55% decrease in suicide attempts and a notable 50% drop in intense suicidal ideation, relative to control groups, 12 months after the interventiona (McGillivray et al., 2020).

In Austraila, a crucial component of the integrated, regionally-based approach to suicide prevention was gatekeeper training, which was widely implemented as a universal approach in secondary schools. Such training programs aimed to equip students with skills to serve as peer gatekeepers, capable of identifying suicide warning signs, addressing concerns, and facilitating appropriate referrals for assistance and care (Mo et al., 2018; Robinson et al., 2018).

The safeTALK, a gatekeeper training initiative, seeks to elevate awareness regarding suicide prevention by framing it as a collective community responsibility, envisioning a helping role for every individual (Turley, 2018). Additionally, it empowers individuals without professional mental health backgrounds to confidently and effectively support someone showing signs of emotional distress. Studies have shown that this training enhances the effectiveness of informal mental health support for those experiencing emotional imbalance. (Kinchin et al., 2020).

Pakistan, located in south-east Asia, grapples with numerous health and social challenges due to persistent waves of violence, political instability, and recurrent changes in the social infrastructure, which has significantly increased the burden of physical and mental ailments impacting individuals of all ages (Hafeez et al., 2023). Unfortunately, Pakistan lacks accurate statistics on suicide deaths and suicidal attempts (Asad & Pirani, 2022), due to under-reporting of such cases, because of social factors, particularly the stigma attached to such cases. However, recently published studies provide some insight into suicide deaths in Pakistan, where adolescents exhibited suicidal ideation and attempts at the rates of 40% and 7%, respectively (Safdar & Afzal, 2021). Moreover, In 2019, suicide mortality rates in Pakistan were estimated to be 8.9 per 100,000 population (Mahesar, Chandio, Latif, Abbas, & Shabbir, 2023; Yasien, Siddiqui, Washdev, & Kumar, 2021). Gilgit-Baltistan (GB) comprising of vallies located among the snow-clad mountains of northern Pakistan, has shown an alarming increase in adolescent mental health issues, including suicidal ideation and suicide rates, which has particularly exacerbated during and following the COVID-19 pandemic (Rahnuma, Fangtong, Khan, Saddique, & Ahmad, 2017).

To address the rising trend of suicidal ideations and attempts, prevention initiatives, such as the safeTALK program hold significance, as they can help in disseminating awareness and education among adolescents through suicide literacy. Programs such as these aim to cultivate courage and confidence among adolescents to openly discuss suicidal thoughts and ideations, and encourage help-seeking behaviors to approach professionals such as psychologists or counselors. Extensive evidence supports the efficacy of the safeTALK program, which has been successfully implemented in various countries (Wilson & Neufeld, 2017). However, Pakistan, with its unique cultural and social setup, has yet to conduct a comprehensive analysis of the effectiveness of such programs.

National and international suicide prevention strategies emphasize the significance of schools for targeted efforts (Brann, Baker, Smith-Millman, Watt, & DiOrio, 2021), as they are conducive and accessible settings for implementing such programs. Leveraging the educational environment effectively enables reach and engagement with adolescents, thereby enabling provision of relevant support and resources to mitigate the risk of suicidal ideation and behavior. Hence, this study intends to validate and assess the effectiveness of RAAHI (guide) and translated and contextualized version, named safeTALK , of the suicide prevention program in GB.

Programs like safeTALK can help lower teen suicides by teaching them about suicide, giving them the confidence to talk about suicidal feelings, and encouraging them to seek help from professionals like psychologists or counselors.

There is sufficient evidence that the safeTALK program is efficient and has been implemented in many other countries (Wilson & Neufeld, 2017). As far as the researcher is aware, Pakistan has never carried out a thorough analysis of the efficacy of such programs. Hence, given the rising suicidal trends in Pakistan, it is crucial to evaluate the contextualized version of safeTALK in addressing this problem of public health importance.

Primary Research Question What is the effect of suicide prevention programs (RAAHI and SafeTALK) in reducing suicidal ideation and in improving mental wellbeing among school-going adolescents in GB? Secondary Research Question

What is the effect of suicide prevention programs (RAAHI and safeTALK) among school going-adolescents in GB on :

1. Suicidal Ideation
2. Suicidal literacy levels
3. Confidence to talk about suicide
4. Willingness to talk about suicide
5. Attitude toward seeking help related to suicidal ideation
6. Depression, Anxiety and Stress level
7. Adaptive coping strategies
8. Self-efficacy Null Hypotheses H01: Suicidal ideation risk among school going-adolescents in GB is similar at baseline and 8-week, following the implementation of the Suicide Prevention Program.

   H02: Compared to baseline, there is no mean difference in suicide literacy, confidence, willingness, and attitude to seek help after 8-week of participation in a Suicide Prevention Program (RAAHI and safeTALK), among school going adolescents.

   H03: Compared to baseline,there is no difference in the mean score of depression, adaptive coping strategies, and self-efficacy after 8-week Suicide Prevention Programs (Raahi and safeTALK)among school-going adolescents METHODS Study Design This research will employ a single group quasi-experimental pre-post interrupted time-series design to allow for examining any change in the levels of the dependent variables before and after the administration of the intervention (Polit & Beck, 2020). Moreover, there will be no control group as it would be unethical to withhold intervention from potentially distressed adolescents (Polit & Beck, 2020).

   Study Phases The study will be carried out in two phases, from January 30, 2024 to October 30, 2024 (Figure 1). Phase I comprised developing 'RAAHI' intervention by the researcher, followed by translation of the safeTALK intervention module, ensuring its contextualization, and validating it through expert review. The effectiveness of the intervention will be evaluated in Phase II using a quasi-experimental pre-post interrupted time-series design. 'RAAHI' focuses on comprehensive suicide literacy and fostering open discussions to combat stigma about suicide, incorporating wellness education, while safeTALK is a shorter, more targeted workshop teaching specific intervention skills and immediate crisis responses using the TALK steps to emphasize immediate practical skills for identifying and addressing suicidal behavior by reducing depression, anxiety and improving adaptive coping strategies and self efficacy level

   Phase IA: Development of the Raahi Module During Phase IA, an interdisciplinary team comprising mental health nurses, psychologists, and educationists will create the RAAHI module for implementation. The objectives, content, timing, and activities for each module will be designed ( Table 1). Experts in the field of mental health will then examine the material for clarity and appropriateness.

   Phase IB: Translation of the safeTALK Intervention Module and Contextual Validation Translation of the Raahi and Safe Talk Interventions material into Urdu, using the backward translation approach, and validation by experts will be carried out to make it culturally and contextually relevant. A team of mental health nurses, clinical psychologists, psychiatrists, and members of the Brain and Mind Institute at the Aga Khan University in Karachi, Pakistan, will validate the intervention module ( Table 1).

   Research Setting GB located in northern Pakistan, boasts spectacular mountain scenery, as it is spread over a region that has two mountain ranges: the Karakoram and Himalayan ranges. Although the region has great natural beauty, it grapples with poverty, limited mental health services, and harsh living conditions. Efforts to improve well-being in GB require addressing these challenges through initiatives. The study will be conducted in four public schools located in northern Pakistan: Diamond Jubilee Model School Daniyore (DJMSD), Daimond Jubilee High School Sonikot (DJHSS), Daimond Jubilee High School Sultanabad (DJHSS) and Daimond Jubilee High School Zulfiqarabad (DJHSZ). The rationale for selecting these schools is chiefly the readiness of the school management to implement, adopt, and sustain the intervention. Since this intervention will be employed in the Pakistani context for the first time, the willingness of the schools principals and their flexibility in mobilizing resources will play a major role. Although the setting will limit external validity, these study sites will be purposively selected, as they will facilitate assessing the feasibility of the intervention in a Pakistani context (Malik & Bi, 2011).

   Study Population Inclusion criteria Both male and female adolescents enrolled in grades IX and X who can comprehend English and Urdu languages will be included. In addition, they and their parents consent to participate in the study.

   Exclusion criterion Adolescents who will be absent or sick on the day of data collection and intervention will not be included in the study.

   Sampling Strategy A multicenter experimental study will be conducted to examine the effectiveness of school-based preventive interventions for suicidal behavior. Using the cluster design, students from four schools in the GB regions will be recruited. The cluster design will ensure inclusivity, as it will enable randomly selecting eligible schools and inviting all students in grades 9 and 10 to participate, preventing discrimination Thee cluster design involves randomizing eligible schools, then recruiting all students of grades 9 and 10, to prevent discrimination. This is the best technique to explore the phenomena and to gain rich data from the participants (Polit & Beck, 2017).

   Sample Size The sample size has been calculated using the G. Power version 3.1.9.2,and Microsoft Excel software using the Paired Sample formula, n = σ²(Z1-β - Z1-α)² / (μ1 - μ2)² and σ² = σ1² - σ2² - 2ρσ1σ2based on the following parameters: A previously published study, conducted by Bailey et al. (2017), reported the mean scores for pre and post-intervention knowledge as 16.88 (16.17 - 17.19) and 20.88 (20.36 - 21.41), respectively, assessment scores (Eleanor Bailey et al., 2020). To convert the standard confidence interval into standard deviation, the following statistical calculation is applied: first, 1.96 is multiplied by 2; then, the t-distribution is used to select the value of 4.128. The standard normal distribution formula has been applied to calculate the SD value. With a 5% statistical significance level, 80% power of the test, and an estimated effect size of 1.2 (Eleanor Bailey et al., 2020), the calculated required sample size was found to be 223 participants.

   Knowledge score

   Mean Confidence interval (95% C.I) Standard limit z-normal at 95% C.I z-value (=2*1.96) Author

   t-distribution

   =tinv (1-0.95,25-1)

   Pre Knowledge assessment score 16.68 16.17 - 17.99 3.92 Bailey, E., et al. (2017). 4.128 2.20446 Post Knowledge assessment score 20.88 20.36 - 21.41 3.92 Bailey, E., et al. (2017). 4.128 1.27180

   To determine the required sample size for a pre-post study, we used the following parameters:
   * Mean difference (μ1 - μ2) =20.16-16.68= 3.84
   * Variance (σ²) = (2.2-1.2)²= 4
   * Desired power (1 - β) = 80%
   * Confidence interval (CI) = 95%
   * Correlation coefficient (ρ) = 0.5 Using the formula for sample size calculation, we plugged in the values and got:n = 222.4 This means that we need a sample size of approximately 223 participants to detect the specified mean difference with the desired level of power and confidence.

   After adding a 20% dropout rate, the final sample size determined is 265 school-going adolescents, who will be recruited for this study.

   Recruitment of Participants Step 1: Participants will be recruited from four schools of Gilgit: Daimond Jubilee Model High School Daniyore (DJMHSD), Daimond Jubilee High School Sonikot (DJHSS), Daimond Jubilee High School Sultanabad (DJHSS) and Daimond Jubilee High School Zulfiqarabad (DJHSZ) through consecutive sampling. After obtaining approval from the concerned school principals, the researcher will meet the administration to request for a teaching room for activity sessions with the adolescents.

   Step 2: A participant flyer will serve as a recruitment tool. Interested students in grades IX and X will be asked to call their parents, for obtaining informed consent, before taking them as research participants.

   Step 3: Parents will be introduced to the study, in a private area. The researcher will discuss the study's procedures and goals, allowing them to ask questions. Obtaining parents' informed consent, which includes permission to assess their child's eligibility for the program, engagement in the intervention, and assessment via pre- and post-testing questionnaires, will be obtained.

   Step 4: Additionally, to ensure compliance with ethical guidelines, a copy of the consent form will also be given to the parents for them to carefully review all the study details. If they agree to allow their children to participate for 30-45 minutes, they will be asked to sign a consent form indicating their consent.

   Step 5: Students will then be assessed for eligibility based on criteria. Participants who meet all eligibility criteria will ultimately be included in the study.

   Procedure Intervention I:"RAAHI" RAAHI is a suicide literacy module that is specially designed to provide individuals with essential knowledge and skills by equipping them with tools to navigate the complexities of mental health and suicide prevention. This module aims to empower people to recognize signs of suicidal ideation, engage in empathetic communication through open discussion, combat stigma, and connect individuals in crisis with appropriate support and resources. The duration of the module will be of three hours. Hence, "RAAHI" seeks to create a world where suicide literacy is widespread, compassion is the key to preventing tragedy, and no one feels isolated in their struggle, thereby contributing to a more empathetic and supportive future (Table 1).

   Intervention II: "safeTALK" The "safeTalk" program is a psychoeducational initiative designed for suicide prevention among adolescents, consisting of a 4-hour workshop that incorporates presentations, videos, discussions, and questions. The workshop is designed according to the standard practices of safeTALK, to assist participants in (a) identifying warning signs of suicide; (b) Avoiding frequent impulses to overlook, dismiss, or avoid discussions about suicide; (c) recognizing and responding to situations where suicidal thoughts may be present by applying fundamental TALK steps (Tell, Ask, Listen, and KeepSafe); and (d) connecting individuals contemplating suicide with first aid assistance and additional community resources (Kinchin et al. (2020). The skills training program concentrates on bolstering adolescents' understanding of activities that promote mental well-being, fostering resilience, honing distress management abilities, and enhancing their capacity to identify early signs of suicidal ideation or behavior, both within themselves and among others. The program also equips participants with strategies for suicide crisis intervention.

   Phase II: Testing the Effectiveness Suicide Prevention Program Pre-Test phase Students willing to participate will be asked to provide their consent, by signing a form/paper, before starting the pen-and-paper pre-training survey. Students will be explicitly informed that participation is entirely voluntary, and their decision to participate or not would not affect their training in any way. First, the psychologist and the researcher will conduct a risk assessment of the students for any prior history or current complaints of suicidal ideation and behavior. A 40-60 minute window will be allocated before the training commences to enable participants to complete the pre-test survey. Additionally, the level of suicidal literacy will also be evaluated through validated and self-report questionnaires. Along with this students' level of confidence and willingness to discuss suicidal ideation and attitudes towards seeking help from others, adopting coping abilities, and self efficacy level will also be assessed. Following the pre-test phase, the students will enter the intervention phase.

   Intervention The intervention phase consists of two workshops, in which the students will be required to participate. The first workshop consists of two hours of "RAAHI intervention", which will provide them general knowledge about suicide, risk factors, consequences, and preventive strategies which will help participants improve their suicide literacy. Moreover, a booklet comprising of different activities will also be provided to participants during the training. Additionally, the second session will introduce the 4-hour safeTALK program, which seeks to increase people's self-awareness and help-seeking behavior, while reducing suicidal ideation. This is a culturally relevant program as it applies basic 'TALK' steps (Tell, Ask, Listen, and KeepSafe); and connects the suicidal person with suicide first aid help and further community resources. Moreover, a pocket card containing the 'suicide alert steps' will also be provided to the participants at the end of the training. In the current study, the safeTALK workshops will be delivered to adolescents, approximately 30 students at a time. The researcher along with a psychologist, will administer this training with the help of translated videos and material in the Urdu language which is culturally appropriate, and has been modified and adapted from the LivingWorks.

   Post-Test phase The data will be re-collected on all outcome measures during post test I, which is right after the intervention, and post test II that will be after 8 weeks of the intervention(Figure 2).

   Data Collection Tools A pre-designed survey will be administered to individuals who express interest in participating in the current study and willingly agree to provide the relevant information. The questionnaire consists of three sections. The first section will gather detailed demographic information and include eligibility questions, followed by the Miller's Modified Scale for Suicidal Ideation (MSSI) (Miller, et al., 1986). Its translated version is available as used in a study of suicide in Pakistan (Andleeb, Ahsan, & Zaheer, 2020). The second section includes questions about suicide literacy, confidence, and willingness to talk abou Time Frame for Data Collection Each participant will receive a short questionnaire at three points in time, labeled as T1, T2 and T3, respectively, as shown in table 1.3. The self-filled questionnaire comprises questions related to suicidal ideation, level of suicidal literacy, level of confidence, and openness to disclose suicidal ideas with others. The researcher will be responsible to look out for missing data and verify them with the participants, wherever it is required and possible. This timely data verification process will enable identifying and correcting the errors present in the data sets.

   Table 2: Time Frame for Data Collection Testing the Effectiveness of Contextually Relevant "Safe Talk" Intervention Pre Intervention (Pre-test Baseline Data): T1 Intervention Immediately Post-intervention I: T2 (Immediate after Intervention) Post- Intervention II: T3 (After 8 weeks)

   Intervention I: Raahi Intervention II: safeTALK

   Data Analysis Data will be entered in a secure, coded format to protect participant anonymity. Statistical analysis will be performed using SPSS version 26. Data normality will be verified. Continuous variables with symmetrical distributions will be summarized using average and standard deviation (SD), while asymmetrical distributions will be described using median and interquartile range (IQR). Categorical variables will be presented with percentages.

   For continuous variables (knowledge, confidence, willingness, and help-seeking), changes over time will be assessed using a linear mixed-effects model. The binary outcome, current suicidal ideation, will be analyzed using a population-averaged generalized estimating equation. Linear regression will estimate beta coefficients and 95% confidence intervals for each predictor variable effect.To compare scores on the suicide literacy scale, repeated measures of ANOVA, with Bonferroni post hoc test, will be calculated, and differences in mean knowledge scores in suicide will be compared.

   Ethical Considerations Researchers must adhere to ethical standards to safeguard research participants, ensuring that their consent is informed and based on a comprehensive understanding of the study. Participation should be voluntary, and the researcher is obligated to uphold confidentiality and anonymity regulations. Hence, the informed consent process will be conducted without coercion or inappropriate influence.

   Ethical approval for the study has been taken from the Ethical Review Committee AKU-ERC (2023-8509-24844) Permission has been taken from the school management. Parents will be invited to the school and the study objectives .will be explained to them. This will provide parents an opportunity to ask questions and give informed consent for participation.

   Informed assent will be taken from students as well, for their participation.Moreover, participants will have a right to withdraw from the study at any time, and in that case, their responses will not be included in the study. All the collected information will be kept confidential. Furthermore, to ensure participant confidentiality, all computer files will be password protected to ensure confidentiality of the data.

   Maintaining anonymity and confidentiality is imperative in the research process. Ensuring anonymity is easy when participant data is detached from their identities. Hence, each participant in this study will be assigned a unique code number and a pseudonym. Additionally, any references to specific health services, doctors, family members, or significant others that could potentially reveal participants' identities will be carefully excluded from the study report.

   Referral Mechanism The data will be collected by trained psychologists and all the identified cases will be referred to a counselor who , will also be hired in the study so he/she can refer the extreme cases for further treatment. The employed counsellors will be on hand at the study sites for data collection and intervention. The cases presenting extreme suicidal ideation thoughts will be referred for follow-up. The screening and referral expenses of the participants will be borne by the study. The attendees will also be informed about the resources that are accessible, such as the hotlines of the suicide prevention organizations operating in Pakistan.

   Potential Risk to Participants The study has no minimal potential risks to the participants. While obtaining informed consent from the parents and assent from the participants, will be made clear that information regarding those considered susceptible, based on their scores, will be shared with their parents and they will be referred for further assessment after parents' consent. However, the status of the participants will be kept confidential from the school authorities. The study will involve psychologists who will conduct this interview along with the principal investigator; hence, they will be able to screen the potential participants.

   Public Health Implications:

   As per the researcher's knowledge, this research study will be the first to establish the effectiveness of a suicide prevention program in improving the mental well-being of school-going adolescents in Pakistan. The results of this research will assist in upscaling contextualized suicide prevention interventions. RAAHI and SafeTALK are expected to bring a positive change in this cohort of adolescents. The success of the intervention will be that people of Pakistan, especially adolescents, start normalizing talking about this taboo topic. This will help to recognize and identify those in need of help in any community. Moreover, awareness regarding suicide may improve resilience and increase help-seeking behavior among adolescents. Ultimately, this preventive intervention program will contribute to reducing the burden of suicide in Pakistan.

   Dissemination The research team plans to share the study findings with the research participants in the Urdu language. Additionally, the results will be communicated to healthcare professionals, and the general public, through the publication of the manuscript in an open-access, peer-reviewed journal, as well as through presentations at various conferences.

   Protocol Amendments Any modifications to the protocol or planned changes will be conveyed to the AKU-ERC-2023-8509-24844, using an online portal.

   Conclusion This study protocol aims to provide crucial insights into the effectiveness of the safeTALK intervention among school-going adolescents in northern Pakistan. The results obtained will serve as a valuable resource for researchers, clinicians, and policymakers, guiding the implementation of more effective suicide prevention strategies tailored to this demographic's need. By assessing the impact of the RAAHI and safeTALK programs on reducing suicidal ideation and enhancing suicide knowledge and confidence levels among participants, over a eight weeks period, this study seeks to share actionable information for improving existing suicide prevention initiatives. The findings from this research hold the potential to influence evidence-based decision-making, supporting the refinement and development of targeted interventions. Ultimately, these efforts aim to contribute to a healthier and more resilient community, by addressing and mitigating the prevalence of suicidal thoughts among adolescents in this region.

   Conflict of Interest None.

ELIGIBILITY:
Inclusion Criteria:

Both male and female adolescents enrolled in grades IX and X who can comprehend English and Urdu languages will be included. In addition, they and their parents consent to participate in the study.

Exclusion Criteria:

Adolescents who will be absent or sick on the day of data collection and intervention will not be included in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — All
Enrollment: 267 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | Pre test, post test I and post test II after 8 weeks
  The degree of suicidal ideation among the participants will be measured through the Modified Scale of Suicidal Ideation by Miller et al. (1991), comprising 21 items. It was translated and used in the Urdu language by Bakht, Saeed, Noushad2, 3, and Shamoon (2017). The MSSI has shown strong internal consistency, with coefficient α ranging from 0.87 to 0.94

SECONDARY OUTCOMES:
Attitude Toward Seeking Professional Psychological Help Scale (ATSPPHS) | Pre test, post test I and post test II after 8 weeks
  5)The Attitude Toward Seeking Professional Psychological Help Scale (ATSPPHS) by Fischer and Farina (1995) will be used to assess participants' attitudes toward seeking help regarding mental health problems. This tool consists of 10 items rated on a Likert scale ranging from 1 (Disagree) to 4 (Agree). The total score, obtained by summing individual item scores, reflects a positive attitude towards seeking psychological help. With reliable psychometric properties, the instrument has a reliability index ranging from 0.80 to 0.86. (Alluhaibi & Awadalla, 2022).
Depression, Anxiety and Stress level. | Pre test, post test I and post test II after 8 weeks
  The Depression, Anxiety, and Stress level will be assessed by DASS-21 questionnaire, which was translated into Urdu, the national language of Pakistan by Bukhari in 2022, to assess the perceived stress levels and psychological well-being of the Pakistani population in Islamabad. Its internal consistency was assessed, revealing a Cronbach's alpha of 0.94. (Gillani, Bukhari, Riaz, & Nisar, 2022). The DASS-21 will serve as a screening tool, evaluating stress, depression, and anxiety over the past week, through 21 items, each consisting of a set of seven questions. Responses on the Likert scale range from 0 to 3, where "never" corresponds to 0, "sometimes" to 1, "frequently" to 2, and "always" to 3. (Beiter et al., 2015). Depression, anxiety, and stress levels of participants will be assessed using predefined cut-off values as follows: depression <6, anxiety <5, and stress <9, in accordance with the DASS-21 guidelines (Gomez, 2016).
Adaptive Coping strategies | Pre test, post test I and post test II after 8 weeks
  7)The Brief-COPE questionnaire, a validated 28-item self-report tool developed.by Carver (1997), assesses both effective and ineffective coping strategies in response to stressful life events. Participants rate their engagement in each strategy on a scale from 1 (not doing at all) to 4 (doing a lot). The questionnaire encompasses of 14 coping including: self-distraction, active coping, denial, substance use, emotional support, instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Scores for each coping style range from 2 to 8, with higher scores indicating a greater inclination towards employing that specific coping mechanism (Salman et al., 2022). The tool has demonstrated a reliability of 0.86 (Ali et al., 2022).

OTHER OUTCOMES:
Self Efficacy | Pre test, post test I and post test II after 8 weeks
  8)Self-efficacy will be measured using a 10-item Generalized Self-Efficacy Scale, which gauges individuals' optimistic beliefs about their personal competence, encompassing determination, problem-solving, and coping skills.(Scholz, Doña, Sud, & Schwarzer, 2002) Responses range from 1 (not at all true) to 4 (exactly true). The urdu translation was already done byMansoor and Ahmad (2022).

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Parpio, PhD, Principal Investigator — Aga Khan University; Rozina Nuruddin, PhD, Study Director — Aga Khan University
Locations (1):
- Aga khan university, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be made publicly available due to privacy concerns and institutional policies. However, the individual participant data (IPD) collected in this study will not be made publicly available due to privacy concerns and institutional policies. The data will be available to researchers upon reasonable request